CLINICAL TRIAL: NCT00950287
Title: Early Detection of Severe Apnea-bradycardia in Preterm Infants Using Algorithm Fusion
Brief Title: Detection of Neonatal Bradycardia
Acronym: INTEM
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2008-A00898-47; PHRC / 08-05 (Other: Rennes University Hospital)
Record Dates: First submitted 2009-07-30; First posted 2009-07-31 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2012-06

CONDITIONS: Apnea; Bradycardia
Keywords: apnea-bradycardias; preterm infants
MeSH Terms: conditions — Apnea; Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cohort: One group of preterm infants
  Interventions: Device: No intervention

INTERVENTIONS:
Device: No intervention — The recordings will be performed in neonatal units with the preterm infant remaining in usual condition with limitations of external stimulation during the study period. The usual monitor will remain in function. The intervention of the nurses in case of apnea will not be modified during the study period. The recording will be obtained from derivation of the signal usually recorded by the monitor in use completed in one centre by a polysomnographic recording (Medtronics France SA), in order to test a possible influence of the sleep status on the detection.

SUMMARY:
Apnea-bradycardia is a frequent phenomenon in preterm infants which has been associated with short term complications and alterations in neurodevelopment. Duration and amplitude of the bradycardias depend on the time delay between the beginning of the bradycardia and the intervention of the nurse.

The purpose of the study is to test a new method set for early detection of bradycardia in preterm infants.

DETAILED DESCRIPTION:
Apnea-bradycardia is a frequent phenomenon in preterm infants which has been associated with short term complications and alterations in neurodevelopment. Duration and amplitude of the bradycardias depend on the time delay between the beginning of the bradycardia and the intervention of the nurse.

The purpose of the study is to test in clinical units and in real life a new method set for early detection of bradycardia in preterm infants.

Each preterm infant cardio-respiratory traces will be recorded during two 4-hours periods of time (the first one at the time of occurrence of apnea-bradycardias and the second one during the following week). During those periods, the alarms of the monitors usually used in the units will also be recorded through automatic detection and these alarms will be compared with the alarms generated by the algorithm tested, for false positive and precocity of the detection. A false positive alarm is a detection which is not associated with a bradycardia of less than 80 bpm. The system will be considered efficient if it allows an earlier detection of severe bradycardias without increasing the number of false positive detection.

ELIGIBILITY:
Inclusion Criteria:

* Parents informed consent
* Presenting with at least 2 significant apnea bradycardia (apnea + decrease in heart rate of more than 33% during at least 4 sec)

Exclusion Criteria:

* Postnatal age of less than 4 days
* Mechanical ventilation
* Severe neurological lesion

Ages: 4 Days to 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants born before 33 weeks of gestational age with a post conceptional age of less than 36 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2009-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Number of false positive alarm detections | 1 week

SECONDARY OUTCOMES:
Delay between the beginning of the bradycardia and the detection. Sensitivity, specificity, positive predictive value, negative predictive value | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Pladys, MD, PhD, Study Director — Rennes University Hospital
Locations (3):
- France (3):
  - Nantes University Hospital, Nantes
  - Rennes University Hospital, Rennes
  - Tours University Hospital, Tours